CLINICAL TRIAL: NCT03427203
Title: Assessment of New Enhanced Ostomy Devices in Real-life Set-tings in Subjects Having an Ileostomy
Brief Title: Assessment of New Ostomy Devices in Subjects Having an Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP264
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): The subjects test the products in the following order
  SenSura Mio (comparator) Coloplast Ostomy device 1 Coloplast Ostomy device 2 Coloplast Ostomy device 3
  Interventions: Device: SenSura Mio; Device: Coloplast Ostomy device 1; Device: Coloplast Ostomy device; Device: Coloplast Ostomy device 3
- Arm 2 (Experimental): The subjects test the products in the following order
  SenSura Mio (comparator) Coloplast Ostomy device 1 Coloplast Ostomy device 3 Coloplast Ostomy device2
  Interventions: Device: SenSura Mio; Device: Coloplast Ostomy device 1; Device: Coloplast Ostomy device; Device: Coloplast Ostomy device 3

INTERVENTIONS:
Device: SenSura Mio — SenSura Mio is a marked ostomy device which is used as the comparator in this study
Device: Coloplast Ostomy device 1 — Coloplast Ostomy device 1 a newly developed ostomy device
Device: Coloplast Ostomy device — Coloplast Ostomy device 2 a newly developed ostomy device
Device: Coloplast Ostomy device 3 — Coloplast Ostomy device 3 a newly developed ostomy device

SUMMARY:
The study investigates the performance of three new adhesives with regard to leakage and the skin condition.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and in DK: signed a letter of authority
2. Be at least 18 years of age and have full legal capacity
3. Have had their ileostomy for at least 3 months
4. Must be able to use custom cut product
5. Can use a product with max cut size 45 mm
6. Self-reported problems with leakage (3 x within 14 days)
7. Get a negative result of a pregnancy test for women of childbearing age (only DK)

Exclusion Criteria:

1. Are currently receiving or have within the past 2 months received radio-and/or chemotherapy (low doses chemotherapy are allowed for other indications than cancer, e.g. below 15 mg methotrexate for rheumatoid arthritis)
2. Are currently receiving or have within the past month received topical steroid treatment in the peristomal skin area, e.g. lotion or spray. Systemic steroid treatment (e.g. injection, or tablet) are allowed.
3. Are pregnant or breastfeeding
4. Are participating in other interventional clinical investigations or have previously participated in this investigation 4.1. Exception: Participation in other Coloplast in-house clinical investigations are accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this (CP264) protocol.
5. Are currently suffering from peristomal skin problems i.e. bleeding and/or broken skin (assessed by the investigator)
6. Have known hypersensitivity towards any of the products used in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 14 days
  Trans epidermal water loss is an objective skin measurement that is measures the evaporation of water on the skin surface using a probe (DermaLab).The trans epidermal water loss is a measure for the skins barrier function. There is always aloss of water from the skin due to evaporation. When the skin barrier is damaged this evaporation of water increases. Thus, transepidermal water loss can be used to assess skin damage

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Medical Director
Locations (3):
- Denmark (2):
  - Coloplast A/S, Humlebæk
  - CCBR Vejle, Vejle
- QPS Netherlands, Groningen, Netherlands